CLINICAL TRIAL: NCT00894803
Title: The "Combined Approach to Lysis Utilizing Eptifibatide and Rt-PA in Acute Ischemic Stroke-Enhanced Regimen" (CLEAR-ER Stroke Trial)
Brief Title: Study of the Combination Therapy of Rt-PA and Eptifibatide to Treat Acute Ischemic Stroke
Acronym: CLEAR-ER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Arthur Pancioli, Dir Academic Med, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P50NS04483-06; 00894803 (Registry Identifier: NCT)
Record Dates: First submitted 2009-05-06; First posted 2009-05-07 (Estimated); Results first posted 2014-03-17 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-03

CONDITIONS: Ischemic Stroke; Stroke; Brain Infarction
Keywords: acute ischemic stroke; stroke; rt-PA, thrombolytic; t-PA; recombinant tissue plasminogen activator; Activase; eptifibatide; Integrilin; fibrinolytic agents; clot dissolving; blood clot
MeSH Terms: conditions — Ischemic Stroke; Stroke; Brain Infarction; Thrombosis | interventions — Eptifibatide; Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rt-PA only (Active Comparator): Subject will receive the standard dose (0.9mg/kg) of IV rt-PA given over 60 minutes. One out of 6 subjects will be in this group.
  Interventions: Drug: rt-PA
- rt-PA and Eptifibatide (Experimental): Subject will receive the standard dose (0.9mg/kg) of IV rt-PA. This IV dose will be discontinued at 40 minutes. The subject will immediately receive an IV bolus of 135mcg/kg eptifibatide followed by an IV infusion of 0.75 mcg/kg/min eptifibatide for 2 hours. Five out of six subjects will be in this group.
  Interventions: Drug: Eptifibatide; Drug: rt-PA

INTERVENTIONS:
Drug: Eptifibatide — IV Eptifibatide is an approved drug by the Food and Drug Administration as a treatment for blood clots causing heart attack and chest pain.Eptifibatide inhibits platelet aggregation by blocking activated platelets from binding fibrinogen.
  Other Names: Integrilin
  Arms: rt-PA and Eptifibatide
Drug: rt-PA — Intravenous recombinant tissue plasminogen activator (rt-PA) is the only approved acute stroke therapy.
  Other Names: Activase

SUMMARY:
The primary goal of this trial is to determine if individuals with acute ischemic stroke treated with a medium dose of IV rt-PA plus IV eptifibatide started within 3 hours of symptom onset are more likely to have a better outcome than individuals treated with standard IV rt-PA alone.

DETAILED DESCRIPTION:
The Combined Approach to Lysis Utilizing Eptifibatide and rt-PA (recombinant tissue plasminogen activator) in Acute Ischemic Stroke-Enhanced Regimen (CLEAR-ER Stroke) trial is a Phase II trial and part of the Specialized Program on Translational Research in Acute Stroke (SPOTRIAS). The overall goals of SPOTRIAS are to enhance delivery of acute stroke patient care and train acute stroke translational researchers.

Stroke most often occurs when blood flow to the brain stops because it is blocked by a blood clot. When a blood clot blocks the blood supply to the brain, parts of the brain may not get enough blood and oxygen to survive. As a result, permanent brain damage can occur, which can affect a person's ability to walk, talk, and function independently. In order to reduce the risk of permanent damage, it is important to restore blood flow to the brain as quickly as possible.

rt-PA, used alone, is already approved by the Food and Drug Administration (FDA) as treatment for patients with a stroke caused by blockage of an artery in the brain and when given within 3 hours of the onset of stroke symptoms. Eptifibatide is also already FDA-approved as a treatment for blood clots causing heart attack. The investigational aspect of this study is the use of eptifibatide for a stroke victim in combination with rt-PA.

The CLEAR Stroke Trial (NCT00250991) demonstrated that the combination of low dose rt-PA plus eptifibatide can be safely given to acute ischemic stroke patients within 3 hours of symptom onset.

The CLEAR-ER Stroke Trial is designed to provide data concerning the risks and benefits of combining eptifibatide with medium dose intravenous rt-PA in 126 acute ischemic stroke patients within 3 hours of symptom onset. Patients will be randomized to a combined intravenous medium-dose rt-PA and eptifibatide regimen, or standard dose rt-PA in a 5 to 1 ratio. This will result in a total of 105 patients treated with a combined regimen, and 21 patients treated with standard dose IV rt-PA alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a serious measurable neurological deficit on the NIH Stroke Scale due to focal brain ischemia.
* An NIH Stroke Scale score >5 at the time the rt-PA is begun.
* Age: 18 through 85 years (i.e. candidates must have had their 18th birthday, but not had their 86th birthday).
* Intravenous rt-PA therapy must be initiated within 3 hours of onset of stroke symptoms.

Exclusion Criteria:

* History of stroke in the past 3 months.
* Previous intra-cranial hemorrhage, neoplasm, subarachnoid hemorrhage, or arterial venous malformation.
* Clinical presentation suggests a subarachnoid hemorrhage, even if initial CT scan is normal.
* Hypertension at time of treatment; systolic BP > 185 or diastolic > 110 mmHg or aggressive measures to lower blood pressure to below these limits are needed.
* Presumed septic embolus.
* Presumed pericarditis including pericarditis after acute myocardial infarction.
* Recent (within 30 days) surgery or biopsy of parenchymal organ.
* Recent (within 30 days) trauma, with internal injuries or ulcerative wounds.
* Recent (within 90 days) severe head trauma or head trauma with loss of consciousness.
* Any active or recent (within 30 days) serious systemic hemorrhage.
* Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency; or oral anticoagulant therapy with Iinternational Normalized Ratio (INR) > 1.7.
* Baseline lab values: positive urine pregnancy test, glucose < 50 or > 400 mg/dl, platelets <100,000 /mm3, Hct (hematocrit) <25 %, or creatinine > 4 mg/dl.
* Ongoing renal dialysis, regardless of creatinine.
* If heparin has been administered within 48 hours, the patient must have a normal partial thromboplastin time (PTT).
* Arterial puncture at a non-compressible site or a lumbar puncture in the previous 7 days.
* Seizure at onset of stroke.
* Pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations.
* Other serious, advanced, or terminal illness or any other condition that the investigator feels would pose a significant hazard to the patient if rt-PA or eptifibatide therapy were initiated.
* Patients whose peripheral venous access is so poor that they are unable to have two standard peripheral intravenous lines started.
* Current participation in another research drug treatment protocol. Patient cannot start another experimental agent until after 90 days.
* Informed consent is not or cannot be obtained.
* Any known history of amyloid angiopathy.
* High density lesion consistent with hemorrhage of any degree.
* Significant mass effect with midline shift.
* Large (more than 1/3 of the middle cerebral artery) regions of clear hypodensity on the baseline CT scan. Sulcal effacement and/or loss of grey-white differentiation alone are not contraindications for treatment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2009-07; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur M Pancioli, MD, Principal Investigator — University of Cincinnati College of Medicine Department of Emergency Medicine; Opeolu M Adeoye, MD, Principal Investigator — University of Cincinnati College of Medicine Department of Emergency Medicine
Locations (20):
- United States (20):
  - UCLA Ronald Reagan Medical Center, Los Angeles, California
  - University of California San Diego, San Diego, California
  - UCLA Medical Center Santa Monica, Santa Monica, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - St. Elizabeth Healthcare Edgewood, Edgewood, Kentucky
  - St. Elizabeth Healthcare Florence, Florence, Kentucky
  - St. Elizabeth Healthcare Ft. Thomas, Fort Thomas, Kentucky
  - Suburban Hospital, Bethesda, Maryland
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Mission Hospital, Inc., Asheville, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - University Hospital, Cincinnati, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio
  - The Jewish Hospital, Cincinnati, Ohio
  - Mercy Hospital, Western Hills, Cincinnati, Ohio
  - Mercy Hospital Mt Airy, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - West Virginia University Hospital, Morgantown, West Virginia

REFERENCES:
- [Background] Barreto AD, Pedroza C, Grotta JC. Adjunctive medical therapies for acute stroke thrombolysis: is there a CLEAR-ER choice? Stroke. 2013 Sep;44(9):2377-9. doi: 10.1161/STROKEAHA.113.001830. Epub 2013 Jul 25. No abstract available. PMID 23887845
- [Result] Pancioli AM, Adeoye O, Schmit PA, Khoury J, Levine SR, Tomsick TA, Sucharew H, Brooks CE, Crocco TJ, Gutmann L, Hemmen TM, Kasner SE, Kleindorfer D, Knight WA, Martini S, McKinney JS, Meurer WJ, Meyer BC, Schneider A, Scott PA, Starkman S, Warach S, Broderick JP; CLEAR-ER Investigators. Combined approach to lysis utilizing eptifibatide and recombinant tissue plasminogen activator in acute ischemic stroke-enhanced regimen stroke trial. Stroke. 2013 Sep;44(9):2381-7. doi: 10.1161/STROKEAHA.113.001059. Epub 2013 Jul 25. PMID 23887841

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in emergency departments at 9 US medical centers comprised of 21 hospitals. Subjects were recruited between July 2009 and October 2012.
Pre-assignment Details: No enrolled participants were excluded from the trial before assignment to groups.
Groups:
- Rt-PA and Eptifibatide: recombinant tissue Plasminogen Activator (rt-PA; 0.6 mg/kg) and Epifibatide (225 mcg/kg)
- Rt-PA Only: recombinant tissue Plasminogen Activator (rt-PA; 0.9 mg/kg)
Period: Overall Study
Arm/Group | Rt-PA and Eptifibatide | Rt-PA Only
Started | 101 | 25
Completed | 81 | 20
Not Completed | 20 | 5
Not completed — Death | 20 | 4
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Rt-PA Only: rt-PA (0.9 mg/kg)
- Rt-PA and Eptifibatide: rt-PA (0.6 mg/kg) and Epifibatide (225 mcg/kg)
- Total: Total of all reporting groups
Arm/Group | Rt-PA Only | Rt-PA and Eptifibatide | Total
Number analyzed (Participants) | 25 | 101 | 126
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 37 | 44
  >=65 years | 18 | 64 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.9 (13.0) | 69.0 (13.6) | 69.3 (13.4)
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 75.5 [60.5 to 81.4] | 71.6 [58.1 to 81.5] | 74.2 [58.1 to 81.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 48 | 60
  Male | 13 | 53 | 66
Region of Enrollment [Number; unit: participants]
  United States | 25 | 101 | 126
National Institutes of Health Stroke Scale Score (NIHSS) [Number; unit: Participants] — National Institutes of Health Stroke Scale Score (NIHSS), 43 point ordinal scale (0 to 42), measuring severity of stroke. 0 (no measurable effect), 42 (dead).
  Participants
    NIHSS <=12 | 10 | 56 | 66
    NIHSS >12 | 15 | 45 | 60
National Institutes of Health Stroke Scale Score (NIHSS) [Mean (Standard Deviation); unit: units on a scale] — National Institutes of Health Stroke Scale Score (NIHSS), 43 point ordinal scale (0 to 42), measuring severity of stroke. 0 (no measurable effect), 42 (dead).
  units on a scale | 16.4 (6.7) | 14.1 (6.9) | 14.6 (6.9)
National Institutes of Health Stroke Scale Score (NIHSS) [Median (Inter-Quartile Range); unit: units on a scale] — National Institutes of Health Stroke Scale Score (NIHSS), 43 point ordinal scale (0 to 42), measuring severity of stroke. 0 (no measurable effect), 42 (dead).
  units on a scale | 17 [11 to 22] | 12 [9 to 20] | 12 [9 to 20]
Stroke symptom onset to intravenous rt-PA start [Number; unit: Participants] — Time from stroke symptom onset to intravenous rt-PA start
  Participants
    < 1 hour | 0 | 1 | 1
    1 to 2 hours | 11 | 56 | 67
    >2 to 3 hours | 13 | 42 | 55
    > 3 hours | 1 | 2 | 3
Stroke symptom onset to intravenous rt-PA start [Median (Inter-Quartile Range); unit: minutes] — Tme from stroke symptom onset to intravenous rt-PA start
  minutes | 129 [90 to 141] | 113 [99 to 135] | 116 [97 to 138]
Modified Rankin Score (mRS) [Number; unit: participants] — modified Rankin Score (mRS), 6 point ordinal scale, measuring functional status. 0 (no symptoms at all), 5 (severe disability; bedridden, incontinent, and requiring constant nursing care)
  participants
    0 | 16 | 74 | 90
    1 | 2 | 11 | 13
    2 | 3 | 7 | 10
    3 | 4 | 4 | 8
    4 | 0 | 5 | 5
    5 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Symptomatic Intracranial Hemorrhage (sICH) Within 36 Hours of Treatment Onset
Description: Primary safety outcome measure - Any ICH related to a decline in neurologic status or the development of new neurologic symptoms which in the judgment of the clinical investigator was related to the ICH. Judgment of significant neurological decline was made by the local clinical investigator
Time Frame: Within 36 hours of initiation of therapy
Measure: Number; unit: participants
Arm/Group | Rt-PA Only | Rt-PA and Eptifibatide
Number analyzed (Participants) | 25 | 101
participants
  sICH within 36 hours of treatment onset | 3 | 2
  No sICH within 36 hours of treatment onset | 22 | 99
Statistical Analysis 1: Comparison: Rt-PA Only vs Rt-PA and Eptifibatide; Test type: Superiority or Other; p = 0.053, Regression, Logistic; an exact logistic regression was used due to the number of events; Odds Ratio (OR) = 0.15, 95% CI 2-sided [0.01 to 1.40] — Arm 2 (rt-PA and Eptifibitide) represents the numerator, Arm 1 (rt-PA only) the denominator

2. Primary Outcome: Modified Rankin Scale (mRS) Score <1 or Return to mRS Baseline
Description: Primary efficacy outcome measure - Modified Rankin Scale of 0 or 1 or return to the pre-stroke value at baseline or better. The scale was performed by a study site investigator not directly involved with acute treatment of the patient. Study subjects dead at 90 days were given a value of '6', and assigned the "bad" outcome. Also those lost to follow-up were assigned the "bad" outcome.
  The Modified Rankin Score (mRS) is a 6 point ordinal scale, measuring functional status. 0 (no symptoms at all), 5 (severe disability; bedridden, incontinent, and requiring constant nursing care).
Time Frame: 90 days from treatment onset
Measure: Number; unit: participants
Arm/Group | Rt-PA Only | Rt-PA and Eptifibatide
Number analyzed (Participants) | 25 | 101
participants
  mRS of 0-1 or return to baseline | 9 | 50
  mRS >1 and > baseline | 16 | 51
Statistical Analysis 1: Comparison: Rt-PA Only vs Rt-PA and Eptifibatide; Test type: Superiority or Other; p = 0.23, Regression, Logistic; Odds Ratio (OR) = 1.74, 95% CI 2-sided [0.70 to 4.31] — Arm 2 (rt-PA and Eptifibitide) represents the numerator, Arm 1 (rt-PA only) the denominator
Statistical Analysis 2: Comparison: Rt-PA Only vs Rt-PA and Eptifibatide; Test type: Superiority or Other; p = 0.53, Regression, Logistic; adjusting for age, baseline NIHSS score and time to IV rt-PA; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.51 to 3.71] — Arm 2 (rt-PA and Eptifibitide) represents the numerator, Arm 1 (rt-PA only) the denominator

3. Other Pre Specified Outcome: Serious Systemic Bleeding
Description: Incidence of serious systemic bleeding defined as requiring transfusion of 2 or more units of packed red blood cells.
Time Frame: Within 7 days of treatment onset
Measure: Number; unit: participants
Arm/Group | Rt-PA Only | Rt-PA and Eptifibatide
Number analyzed (Participants) | 25 | 101
participants
  Serious systemic bleeding | 0 | 1
  No Serious systemic bleeding | 25 | 100

4. Other Pre Specified Outcome: Symptomatic Intracranial Hemorrhage (sICH) Within 7 Days of Treatment Onset
Description: Any ICH related to a decline in neurologic status or the development of new neurologic symptoms which in the judgment of the clinical investigator was related to the ICH. Judgment of significant neurological decline was made by the local clinical investigator
Time Frame: Within 7 days of treatment onset
Measure: Number; unit: participants
Arm/Group | Rt-PA Only | Rt-PA and Eptifibatide
Number analyzed (Participants) | 25 | 101
participants
  sICH within 7 days of treatment onset | 3 | 2
  No sICH within 7 days of treatment onset | 22 | 99
Statistical Analysis 1: Comparison: Rt-PA Only vs Rt-PA and Eptifibatide; Test type: Superiority or Other; p = 0.053, Regression, Logistic; Exact method used due to number of responses; Odds Ratio (OR) = 0.15, 95% CI 2-sided [0.01 to 1.40] — Arm 2 (rt-PA and Eptifibitide) represents the numerator, Arm 1 (rt-PA only) the denominator

5. Other Pre Specified Outcome: Asymptomatic Intracranial Hemorrhage (asICH) Within 7 Days of Treatment Onset
Description: Any ICH observed on CT by the study site neuroradiologist and the independent study neuroradiologist; the central reader. The ICH would not be related to a decline in neurologic status or the development of new neurologic symptoms which in the judgment of the clinical investigator was related to the ICH,where judgment of significant neurological decline was made by the local clinical investigator. A third independent reader will make the final determination if there is disagreement between the treating investigator and the central reader
Time Frame: Within 7 days of treatment onset
Measure: Number; unit: participants
Arm/Group | Rt-PA Only | Rt-PA and Eptifibatide
Number analyzed (Participants) | 25 | 101
participants
  asICH within 7 days of treatment onset | 3 | 16
  No asICH within 7 days of treatment onset | 22 | 85
Statistical Analysis 1: Comparison: Rt-PA Only vs Rt-PA and Eptifibatide; Test type: Superiority or Other; p = 0.76, Regression, Logistic; Odds Ratio (OR) = 1.38, 95% CI [0.35 to 8.02] — Arm 2 (rt-PA and Eptifibitide) represents the numerator, Arm 1 (rt-PA only) the denominator

6. Other Pre Specified Outcome: Death Within 7 Days of Treatment Onset
Description: Death due to any cause within 7 days of treatment onset
Time Frame: Within 7 days of treatment onset
Measure: Number; unit: participants
Arm/Group | Rt-PA Only | Rt-PA and Eptifibatide
Number analyzed (Participants) | 25 | 101
participants
  Death within 7 days of treatment onset | 3 | 12
  No death within 7 days of treatment onset | 22 | 89
Statistical Analysis 1: Comparison: Rt-PA Only vs Rt-PA and Eptifibatide; Test type: Superiority or Other; p = 0.99999, Regression, Logistic; Exact method used due to small number of responses; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.24 to 5.92] — Arm 2 (rt-PA and Eptifibitide) represents the numerator, Arm 1 (rt-PA only) the denominator

7. Other Pre Specified Outcome: Death Due to Stroke Within 7 Days of Treatment Onset
Description: Death due to stroke within 7 days of treatment onset. Classified by blinded clinical investigators
Time Frame: Within 7 days of treatment onset
Measure: Number; unit: participants
Arm/Group | Rt-PA Only | Rt-PA and Eptifibatide
Number analyzed (Participants) | 25 | 101
participants
  Death due to stroke within 7 days of treatment ons | 3 | 12
  No Death due to stroke within 7 days of treatment | 22 | 89
Statistical Analysis 1: Comparison: Rt-PA Only vs Rt-PA and Eptifibatide; Test type: Superiority or Other; p = 0.99999, Regression, Logistic; Exact method used due to number of responses; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.24 to 5.92] — Arm 2 (rt-PA and Eptifibitide) represents the numerator, Arm 1 (rt-PA only) the denominator

8. Post Hoc Outcome: Death Within 90 Days of Treatment Onset
Description: Death due to any cause within 90 days of treatment onset
Time Frame: Within 90 days of treatment onset
Measure: Number; unit: participants
Arm/Group | Rt-PA Only | Rt-PA and Eptifibatide
Number analyzed (Participants) | 25 | 101
participants
  Death within 90 days of treatment onset | 4 | 20
  No death within 90 days of treatment onset | 21 | 81
Statistical Analysis 1: Comparison: Rt-PA Only vs Rt-PA and Eptifibatide; Test type: Superiority or Other; p = 0.78, Regression, Logistic; Exact methods used due t number of responses; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.38 to 5.76] — Arm 2 (rt-PA and Eptifibitide) represents the numerator, Arm 1 (rt-PA only) the denominator

9. Post Hoc Outcome: Death Due to Stroke Within 90 Days of Treatment Onset
Description: Death due to stroke within 90 days of treatment onset. Classified by blinded clinical investigators
Time Frame: Within 90 days of treatment onset
Measure: Number; unit: participants
Arm/Group | Rt-PA Only | Rt-PA and Eptifibatide
Number analyzed (Participants) | 25 | 101
participants
  Death due to stroke within 90 days of treatment on | 4 | 15
  No Death due to stroke within 90 days of treatment | 21 | 86
Statistical Analysis 1: Comparison: Rt-PA Only vs Rt-PA and Eptifibatide; Test type: Superiority or Other; p = 0.99999, Regression, Logistic; Exact method used due to number of responses; Odds Ratio (OR) = .92, 95% CI 2-sided [0.26 to 4.18] — Arm 2 (rt-PA and Eptifibitide) represents the numerator, Arm 1 (rt-PA only) the denominator

10. Secondary Outcome: Barthel Index ≥ 95
Description: Barthel index score of ≥ 95. The scale was performed by a study site investigator not directly involved with acute treatment of the patient. Study subjects dead at 90 days and those lost to follow-up were assigned the "bad" outcome.
  The Barthel index is a score comprised of 10 individual items. Each item may be scored 0, 5, 10 or 15; not all items use the full range of 4 possible values. The individual items are summed to produce a total score between 0 and 100; where 0 is inferior performance and 100 is optimal. A score of ≥ 95 is usually considered excellent.
Time Frame: 90 days from treatment onset
Measure: Number; unit: participants
Arm/Group | Rt-PA Only | Rt-PA and Eptifibatide
Number analyzed (Participants) | 25 | 101
participants
  Barthel Index ≥ 95 | 11 | 55
  Barthel Index < 95 | 14 | 46
Statistical Analysis 1: Comparison: Rt-PA Only vs Rt-PA and Eptifibatide; Test type: Superiority or Other; p = 0.35, Regression, Logistic; Odds Ratio (OR) = 1.52, 95% CI 2-sided [0.63 to 3.67] — Arm 2 (rt-PA and Eptifibitide) represents the numerator, Arm 1 (rt-PA only) the denominator
Statistical Analysis 2: Comparison: Rt-PA Only vs Rt-PA and Eptifibatide; Test type: Superiority or Other; p = 0.85, Regression, Logistic; adjusting for age, baseline NIHSS and time to IV rt-PA; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.40 to 3.02] — Arm 2 (rt-PA and Eptifibitide) represents the numerator, Arm 1 (rt-PA only) the denominator

11. Secondary Outcome: Glasgow Outcome Scale (GOS) of 1
Description: Glasgow outcome scale score of 1 versus greater than 1. The scale was performed by a study site investigator not directly involved with acute treatment of the patient. Study subjects dead at 90 days and those lost to follow-up were assigned the "bad" outcome.
  The Glasgow Outcome Scale is scored; 1=good recovery, 2=moderately disabled, 3=severely disabled, 4=vegetative survival, 5=dead.
Time Frame: 90 days from treatment onset
Measure: Number; unit: participants
Arm/Group | Rt-PA Only | Rt-PA and Eptifibatide
Number analyzed (Participants) | 25 | 101
participants
  GOS =1 | 10 | 52
  GOS > 1 | 15 | 49
Statistical Analysis 1: Comparison: Rt-PA Only vs Rt-PA and Eptifibatide; Test type: Superiority or Other; p = 0.30, Regression, Logistic; Odds Ratio (OR) = 1.59, 95% CI 2-sided [0.65 to 3.88] — Arm 2 (rt-PA and Eptifibitide) represents the numerator, Arm 1 (rt-PA only) the denominator
Statistical Analysis 2: Comparison: Rt-PA Only vs Rt-PA and Eptifibatide; Test type: Superiority or Other; p = 0.73, Regression, Logistic; adjusting for age, baseline NIHSS and time to IV rt-PA; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.44 to 3.24] — Arm 2 (rt-PA and Eptifibitide) represents the numerator, Arm 1 (rt-PA only) the denominator

12. Other Pre Specified Outcome: NIH Stroke Scale Score (NIHSS) ≤ 5
Description: Study subjects with an NIH stroke scale score of ≤ 5 at 2 hours from treatment onset, those sedated and unable to be evaluated by the NIHSS were assigned the "bad" outcome (n=1).
  The NIH stroke scale score is scale based on 15 items individually scored between 0-2, 0-3 or 0-4 depending upon the item. The individual items are summed to produce a score between 0 and 42, where 0 indicates no deficit and 42 indicates death.
Time Frame: Within 2 hours of treatment onset
Measure: Number; unit: participants
Arm/Group | Rt-PA Only | Rt-PA and Eptifibatide
Number analyzed (Participants) | 25 | 101
participants
  NIHSS ≤ 5 | 6 | 35
  NIHSS > 5 | 19 | 66
Statistical Analysis 1: Comparison: Rt-PA Only vs Rt-PA and Eptifibatide; Test type: Superiority or Other; p = 0.31, Regression, Logistic; Odds Ratio (OR) = 1.68, 95% CI 2-sided [0.61 to 4.99] — Arm 2 (rt-PA and Eptifibitide) represents the numerator, Arm 1 (rt-PA only) the denominator

13. Other Pre Specified Outcome: NIH Stroke Scale Score (NIHSS) ≤ 2
Description: Study subjects with an NIH stroke scale score of ≤ 2 at 24 hours from treatment onset, those dead (n=1) or sedated and unable to be evaluated by the NIHSS were assigned the "bad" outcome (n=5).
  The NIH stroke scale score is scale based on 15 items individually scored between 0-2, 0-3 or 0-4 depending upon the item. The individual items are summed to produce a score between 0 and 42, where 0 indicates no deficit and 42 indicates death.
Time Frame: Within 24 hours of treatment onset
Measure: Number; unit: participants
Arm/Group | Rt-PA Only | Rt-PA and Eptifibatide
Number analyzed (Participants) | 25 | 101
participants
  NIHSS ≤ 2 | 5 | 27
  NIHSS > 2 | 20 | 74
Statistical Analysis 1: Comparison: Rt-PA Only vs Rt-PA and Eptifibatide; Test type: Superiority or Other; p = 0.55, Regression, Logistic; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.47 to 4.07] — Arm 2 (rt-PA and Eptifibitide) represents the numerator, Arm 1 (rt-PA only) the denominator

14. Other Pre Specified Outcome: NIH Stroke Scale Score (NIHSS) ≤2 at 90 Days
Description: Study subjects with an NIH stroke scale score ≤ 2 points at 90 days from treatment onset compared to baseline value, those dead or unable to be evaluated by the NIHSS were assigned the "bad" outcome.
  The NIH stroke scale score is scale based on 15 items individually scored between 0-2, 0-3 or 0-4 depending upon the item. The individual items are summed to produce a score between 0 and 42, where 0 indicates no deficit and 42 indicates death.
Time Frame: 90 days from treatment onset
Measure: Number; unit: participants
Arm/Group | Rt-PA Only | Rt-PA and Eptifibatide
Number analyzed (Participants) | 25 | 101
participants
  NIHSS ≤ 2 | 11 | 45
  NIHSS > 2 | 14 | 56
Statistical Analysis 1: Comparison: Rt-PA Only vs Rt-PA and Eptifibatide; Test type: Superiority or Other; p = 0.82, Regression, Logistic; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.46 to 2.67] — Arm 2 (rt-PA and Eptifibitide) represents the numerator, Arm 1 (rt-PA only) the denominator

15. Post Hoc Outcome: Modified Rankin Scale (mRS) of 0-1
Description: Modified Rankin Scale of 0 or 1. The scale was performed by a study site investigator not directly involved with acute treatment of the patient. Study subjects dead at 90 days were given a value of '6', and assigned the "bad" outcome. Also those lost to follow-up were assigned the "bad" outcome.
  The Modified Rankin Score (mRS) is a 6 point ordinal scale, measuring functional status. 0 (no symptoms at all), 5 (severe disability; bedridden, incontinent, and requiring constant nursing care).
Time Frame: 90 days from treatment onset
Measure: Number; unit: participants
Arm/Group | Rt-PA Only | Rt-PA and Eptifibatide
Number analyzed (Participants) | 25 | 101
participants
  mRS of 0-1 | 6 | 44
  mRS > 1 | 19 | 57
Statistical Analysis 1: Comparison: Rt-PA Only vs Rt-PA and Eptifibatide; Test type: Superiority or Other; p = 0.07, Regression, Logistic; Odds Ratio (OR) = 2.44, 95% CI 2-sided [0.90 to 6.64] — Arm 2 (rt-PA and Eptifibitide) represents the numerator, Arm 1 (rt-PA only) the denominator
Statistical Analysis 2: Comparison: Rt-PA Only vs Rt-PA and Eptifibatide; Test type: Superiority or Other; p = 0.22, Regression, Logistic; adjusting for age, baseline NIHSS and time to IV rt-PA; Odds Ratio (OR) = 1.98, 95% CI 2-sided [0.67 to 5.88] — Arm 2 (rt-PA and Eptifibitide) represents the numerator, Arm 1 (rt-PA only) the denominator

ADVERSE EVENTS:
Time Frame: Up to 90 days from initiation of therapy
Description: Adverse events were documented as recorded in the medical record until discharge. The occurrence of adverse events from the time of hospital discharge to the 90 day visit was collected at the time of the 90 day visit.
Arm/Group | Rt-PA Only | Rt-PA and Eptifibatide
Serious Adverse Events (participants affected / at risk) | 7/25 | 26/101
Other Adverse Events (participants affected / at risk) | 17/25 | 80/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rt-PA Only (N=25) | Rt-PA and Eptifibatide (N=101)
Anaemias nonhaemolytic and marrow depression (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arteriosclerosis, stenosis, vascular insufficiency and necrosis (Vascular disorders) | 1 (1) | 3 (3)
Cardiac therapeutic procedures (Surgical and medical procedures) | 0 (0) | 1 (1)
Central nervous system vascular disorders (Nervous system disorders) | 1 (1) | 1 (1)
Communication disorders and disturbances (Psychiatric disorders) | 1 (1) | 0 (0)
Coronary artery disorders (Cardiac disorders) | 0 (0) | 3 (3)
Deliria (incl confusion) (Psychiatric disorders) | 0 (0) | 1 (1)
Embolism and thrombosis (Vascular disorders) | 2 (2) | 2 (2)
Gallbladder disorders (Hepatobiliary disorders) | 0 (0) | 2 (2)
Gastrointestinal haemorrhages NEC (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastrointestinal inflammatory conditions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal signs and symptoms (Gastrointestinal disorders) | 1 (1) | 0 (0)
General system disorders NEC (General disorders) | 0 (0) | 1 (1)
Genitourinary tract disorders NEC (Renal and urinary disorders) | 0 (0) | 1 (1)
Heart failures (Cardiac disorders) | 0 (0) | 1 (1)
Increased intracranial pressure and hydrocephalus (Nervous system disorders) | 0 (0) | 5 (5)
Infections - pathogen unspecified (Infections and infestations) | 0 (0) | 5 (5)
Injuries NEC (Injury, poisoning and procedural complications) | 0 (0) | 5 (5)
Muscle disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neurological disorders NEC (Nervous system disorders) | 2 (3) | 3 (3)
Neuromuscular disorders (Nervous system disorders) | 1 (1) | 0 (0)
Pulmonary vascular disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Renal disorders (excl nephropathies) (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory disorders NEC (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Respiratory tract infections (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Seizures (incl subtypes) (Nervous system disorders) | 0 (0) | 1 (1)
Vascular haemorrhagic disorders (Vascular disorders) | 1 (1) | 3 (3)
Vascular therapeutic procedures (Surgical and medical procedures) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rt-PA Only (N=25) | Rt-PA and Eptifibatide (N=101)
Administration site reactions (General disorders) | 0 (0) | 5 (6)
Administration site reactions (Injury, poisoning and procedural complications) | 0 (0) | 5 (5)
Allergic conditions (Immune system disorders) | 0 (0) | 5 (5)
Anaemias nonhaemolytic and marrow depression (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Angioedema and urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)
Anxiety disorders and symptoms (Psychiatric disorders) | 2 (2) | 4 (4)
Arteriosclerosis, stenosis, vascular insufficiency and necrosis (Vascular disorders) | 0 (0) | 2 (2)
Bacterial infectious disorders (Infections and infestations) | 1 (2) | 0 (0)
Body temperature conditions (General disorders) | 3 (3) | 7 (7)
Bone, calcium, magnesium and phosphorus metabolism disorders (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
Bronchial disorders (excl neoplasms) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cardiac arrhythmias (Cardiac disorders) | 5 (5) | 8 (9)
Cardiac disorder signs and symptoms (Cardiac disorders) | 0 (0) | 3 (4)
Central nervous system vascular disorders (Nervous system disorders) | 0 (0) | 2 (2)
Changes in physical activity (Psychiatric disorders) | 0 (0) | 1 (1)
Cognitive and attention disorders and disturbances (Psychiatric disorders) | 0 (0) | 1 (1)
Coronary artery disorders (Cardiac disorders) | 1 (1) | 1 (1)
Decreased and nonspecific blood pressure disorders and shock (Vascular disorders) | 2 (2) | 4 (4)
Dental and gingival conditions (Gastrointestinal disorders) | 0 (0) | 3 (3)
Depressed mood disorders and disturbances (Psychiatric disorders) | 0 (0) | 1 (1)
Device issues (General disorders) | 0 (0) | 1 (1)
Electrolyte and fluid balance conditions (Metabolism and nutrition disorders) | 3 (3) | 16 (16)
Embolism and thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Enzyme investigations NEC (Investigations) | 1 (1) | 0 (0)
Epidermal and dermal conditions (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)
Eye disorders NEC (Eye disorders) | 0 (0) | 1 (1)
Fungal infectious disorders (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal motility and defaecation conditions (Gastrointestinal disorders) | 1 (1) | 9 (9)
Gastrointestinal signs and symptoms (General disorders) | 7 (7) | 15 (22)
General system disorders NEC (General disorders) | 4 (4) | 5 (5)
Genitourinary tract disorders NEC (Renal and urinary disorders) | 4 (4) | 7 (7)
Glucose metabolism disorders (incl diabetes mellitus) (Endocrine disorders) | 0 (0) | 4 (4)
Glucose metabolism disorders (incl diabetes mellitus) (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Haematology investigations (incl blood groups) (Investigations) | 1 (1) | 1 (1)
Headaches (Nervous system disorders) | 4 (4) | 21 (21)
Heart failures (Cardiac disorders) | 2 (2) | 0 (0)
Increased intracranial pressure and hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Infections - pathogen unspecified (Infections and infestations) | 3 (3) | 10 (10)
Injuries NEC (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Joint disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Lower respiratory tract disorders (excl obstruction and infection) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Muscle disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal and connective tissue disorders NEC (Musculoskeletal and connective tissue disorders) | 1 (1) | 12 (14)
Neurological disorders NEC (Nervous system disorders) | 5 (5) | 11 (11)
Neuromuscular disorders (Nervous system disorders) | 0 (0) | 3 (3)
Penile and scrotal disorders (excl infections and inflammations) (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Physical examination and organ system status topics (Investigations) | 0 (0) | 1 (1)
Pleural disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Procedural related injuries and complications NEC (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Renal disorders (excl nephropathies) (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory disorders NEC (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (10)
Respiratory tract infections (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Seizures (incl subtypes) (Nervous system disorders) | 1 (1) | 1 (1)
Sleep disorders and disturbances (Psychiatric disorders) | 0 (0) | 2 (2)
Sleep disturbances (incl subtypes) (Nervous system disorders) | 0 (0) | 2 (2)
Tongue conditions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract disorders (excl infections) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Urinary tract signs and symptoms (Renal and urinary disorders) | 2 (2) | 5 (5)
Urolithiases (Renal and urinary disorders) | 0 (0) | 1 (1)
Vascular haemorrhagic disorders (Vascular disorders) | 0 (0) | 12 (16)
Water, electrolyte and mineral investigations (Investigations) | 0 (0) | 1 (1)
White blood cell disorders (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes